CLINICAL TRIAL: NCT07032623
Title: Neuromuscular Effects of Spinal Manipulation in Individuals Following Anterior Cruciate Ligament Reconstruction: A Single-Blinded Randomized Controlled Trial
Brief Title: Neuromuscular Effects of Spinal Manipulation in Individuals Following Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Ricardo Paredes, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 070520243082024
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Knee; Anterior cruciate ligament; Motor control; Electromyography; Physiotherapy
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Spinal Manipulation (Experimental)
  Interventions: Procedure: Spinal Manipulation

INTERVENTIONS:
Procedure: Spinal Manipulation — The spinal manipulation will target the sacroiliac joint using the global pelvic manipulation technique. Participants will be positioned in lateral decubitus with the ACL-reconstructed limb placed uppermost. The therapist will apply progressive rotation and flexion at the hip and knee joints to increase tissue tension. To establish contact, the therapist's knee will be placed against the participant's flexed knee. A high-velocity, low-amplitude thrust will then be delivered to optimize joint motion, with cavitation being monitored throughout the procedure.
  Arms: Spinal Manipulation

SUMMARY:
This single-blind, randomized controlled trial aims to investigate the effects of spinal manipulation on neuromuscular control in individuals with anterior cruciate ligament reconstruction during a single-leg vertical drop landing task. The intervention group will receive spinal manipulation, while the control group will not receive any therapeutic intervention. The main question it aims to answer is:

• Can spinal manipulation induce changes in muscle activation, co-contraction magnitude, and biomechanical parameters during landing?

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone anterior cruciate ligament reconstruction
* Successful return to recreational sports participation

Exclusion Criteria:

* Peripheral or central neurological disorders
* Systemic or degenerative diseases
* History of spinal surgery
* Contraindications to spinal manipulation
* Low back or sacroiliac pain within the previous month
* Prior exposure to manipulative therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Co-contraction Index | Outcome measures will be assessed at baseline and 10 minutes post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rehabilitation Research (CIR), School of Health of Polytechnic of Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided